CLINICAL TRIAL: NCT03622684
Title: Progressive Muscle Relaxation According to Jacobson in Treatment of the Patients With Temporomandibular Joint Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Ewa Ferendiuk, MD, Doctor of medical sciences, assistant, research worker, principal investigator of Jagiellonian University, Medical College, Prosthodontic Department, Room of Functional Disorders of Masticatory System, Poland, Krakow, Jagiellonian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBET/192/B/2013
Record Dates: First submitted 2017-11-21; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: TEMPOROMANDIBULAR JOINT DYSFUNCTION SYNDROME
Keywords: TMJ- temporomandibular joint-disorder; Muscle relaxation; Psychoemotional factor; Stress
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle relaxation according to Jacobson (Experimental): . Does the use of the method of progressive relaxation according to Jacobson will be beneficial to reduce pain and improve the functioning of the stomatognathic system being evaluated in clinical trials?
  Interventions: Behavioral: Muscle relaxation according to Jacobson

INTERVENTIONS:
Behavioral: Muscle relaxation according to Jacobson

SUMMARY:
Temporomandibular joint disorders are ranked third among the most common stomatological diseases after dental caries and periodontal problems. Type of dysfunction is determined by environmental, genetic and psycho-emotional factors. It has been observed that increasing level of stress leads to the increase of harmful parafunctional habits in the stomatognathic system whose long-term effect prevents the ability of the organism to compensate and adapt the function, which contributes to the pain within the masticatory system. Nowadays applied methods in treatment of temporomandibular joint disorders are still under investigation. However, they have not been developed effectively yet. Satisfactory methods of masticatory muscle relaxation (with the exception for drug treatment) are only related to mental patients. Significant impact factor and psycho-emotional stress in the etiology of dysfunction indicate the need of the routine approach in the treatment of patients with temporomandibular joint disorders to be changed. The attempt to cooperate with a psychologist may facilitate the effectiveness of traditional rehabilitation of patients with dysfunction.

DETAILED DESCRIPTION:
Introduction In the 30s of the previous century, Edmund Jacobson developed the method of progressive muscle relaxation, which is based on the premise that mental relaxation should naturally result from physical relaxation. The primary objective of Jacobson's relaxation is to increase patient's awareness associated with the feeling of muscle tension, no matter how intense it is. This method teaches patients how to take control over the factors causing stress, with simultaneous relaxation of skeletal muscles, and alternating tension and relaxation deliberately in the next group of striated muscle. Regular training is aimed at developing a habit of locating the tension and loosening individual muscle groups. Data from the literature indicates the usefulness of Jacobson's progressive muscle relaxation method as a supportive therapy for the treatment of neurological disorders, depression, anxiety, bronchial asthma, and cardiological conditions. Positive therapeutic results have also been reported in the treatment of peptic ulcer, chronic headache, tinnitus, sleep disorders, and psychological treatment of neurological conditions. The additional benefits of this therapeutic approach include reduced anxiety, decreased arterial hypertension and improved heart function, improved gastric and intestinal function, increased imagination and thought processes, increased trust between the patient and the physician, and improved control of one's mood. Jacobson's progressive muscle relaxation has not been used in the treatment of temporomandibular joint disorders. The above has become an inspiration to undertake research in this field. The significant impact of psycho-emotional factors and stress on the rise or worsening of dysfunction as well as cooperation with the psychologist can significantly influence the course and treatment of functional disorders. The elimination of psychological components in patients with temporomandibular joint disorders may contribute to the reduction of pain and frequency of parafunctional habits.

The aim of the study was to obtain data, documented test results as to the efficiency of progressive muscle relaxation in the treatment of pain caused by temporomandibular joint disorders, as a supplement to previous methods using occlusal splint and other physical therapies. The study also included the treatment of post-isometric muscle relaxation. In order to ensure an objective comparative evaluation of these two methods of adjunctive treatment, clinical studies and surveys were conducted. The aim of the study was to answer the following questions:

1. Does the use of Jacobson's progressive relaxation method will be beneficial to reduce pain and improve the functioning of the stomatognathic system being evaluated in clinical trials?
2. Does the relaxation method obtain a positive opinion of the patients and can complement the previously used prosthetic rehabilitation with occlusal splint as well as other physical therapies?
3. Which one of assessed methods (progressive muscle relaxation according to Jacobson and method of post- isometric relaxation) gains an advantage in the treatment used in the adjunctive therapy of temporomandibular joint disorders, and assessment of which according to their impact on muscle relaxation on the basis of the clinical trial and the results of the survey? Material and Methods The study included 100 patients of both sexes, aged from 20 to 35 years who were diagnosed with pain due to temporomandibular joint disorders accompanied with high muscle tension of masticatory muscles. The study included patients reported to prosthetic treatment to Department of Prosthodontics at the Jagiellonian University, Medical College in Krakow between 2014 and 2016. Patients were divided into two groups of 50 people each. In the group number I-test group, treatment was performed by progressive muscle relaxation according to Jacobson. In the group number II- control group, post-isometric muscle relaxation treatment was instituted. The following criteria the patients had to meet in order to be included in the study: good general health, painful form of temporomandibular joint disorders with high muscle tension, pain lasting for at least 3 weeks prior to admission, and also patients with full arches without previous orthodontic treatment.

The exclusion criteria included: joint component of functional disorders (pain in the temporomandibular joints, acoustic symptoms), deterioration of the posture resulting from relaxation training (aggravation of muscular pain, worsening of mental state) unstable musculoskeletal system (frequent painful muscle spasms), tetanus, other diseases that prevent the patient from continuing the study (fever), and the lack of the patient's informed consent.

The criterion for the allocation of patients to groups I and II was the consent to perform relaxation treatments for the treatment of functional disorders of the chewing organ and the lack of contraindications.

Relaxation therapy schedule was adapted to clinical and laboratory stages of occlusion splint. For the purposes of the research both physiotherapy and pharmacological treatment were eliminated. Following the purpose of the studies, comparative evaluation of two supporting methods of treatment were undertaken: for the patients with temporomandibular joint disorders, the performance of 5 cycles of progressive muscle relaxation according to Jacobson in the group I - the study one, and 5 cycles of post- isometric muscle relaxation in group II - control. The qualification and assignment of the patients into group I and II were based on the results of clinical and specialist examination. In group I the training was held twice a week and was conducted by a qualified psychologist. Each meeting lasted 45 minutes. The procedure was to tighten the subsequent muscle groups for 5-7 seconds, followed by a 20-second relaxation time. The basic part of the training performed during the first two meetings included alternating tension and relaxation of muscles in the limbs, abdomen and face based on Jacobson's classic training. The next session was modified taking into account the muscles of the neck and face, and the fourth and fifth sessions included exercises with which the patient was familiarized during earlier training, but done separately for each part of the face.In group II the treatment was conducted by a qualified physiotherapist and also was held twice a week, 45 minutes each, and next exercises were repeated three times.

ELIGIBILITY:
Inclusion Criteria:

1. good general health
2. painful form of temporomandibular joint disorders- masticatory muscles pain with high muscle tension
3. pain lasting for at least 3 weeks prior to admission
4. patients with full arches without previous orthodontic treatment.

Exclusion Criteria:

1. joint component of functional disorders (pain in the temporomandibular joints, acoustic symptoms)
2. deterioration of the posture resulting from relaxation training (aggravation of muscular pain, worsening of mental state)
3. unstable musculoskeletal system (frequent painful muscle spasms), tetanus, other diseases that prevent the patient from continuing the study (fever)
4. the lack of the patient's informed consent.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study included 100 patients of both sexes, aged from 20 to 35 years who were diagnosed with pain due to temporomandibular joint disorders accompanied with high muscle tension of masticatory muscles.
Enrollment: 100 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with assesment of psycho emotional factor and stress | 2 years
  Analyses based on a survey questionnaire in the development of their own - scoring scale

SECONDARY OUTCOMES:
Incidence of CIB values in both groups before and after treatments relaxation assessed by specialized statistical package "R" i386 | 1 Month
  The results of the research were obtained using specialized statistical package "R" i386 3.2.3. To check the theoretical dependence (hypothesis testing), Chi-square test of Pearson was used. To compare the relationship between the results obtained in clinical trials (comparison between the two dependent samples), Anova parametric test was performed.The specific results of research were presented in tables and figures.
Incidence of OBC values in both groups before and after treatments relaxation assessed by specialized statistical package "R" i386 | 1 Month
  The results of the research were obtained using specialized statistical package "R" i386 3.2.3. To check the theoretical dependence (hypothesis testing), Chi-square test of Pearson was used. To compare the relationship between the results obtained in clinical trials (comparison between the two dependent samples), Anova parametric test was performed.The specific results of research were presented in tables and figures.

REFERENCES:
- [Background] Alvarez-Arenal A, Junquera LM, Fernandez JP, Gonzalez I, Olay S. Effect of occlusal splint and transcutaneous electric nerve stimulation on the signs and symptoms of temporomandibular disorders in patients with bruxism. J Oral Rehabil. 2002 Sep;29(9):858-63. doi: 10.1046/j.1365-2842.2002.00923.x. PMID 12366541
- [Background] Almoznino G, Zini A, Zakuto A, Sharav Y, Haviv Y, Hadad A, Chweidan H, Yarom N, Benoliel R. Oral Health-Related Quality of Life in Patients with Temporomandibular Disorders. J Oral Facial Pain Headache. 2015 Summer;29(3):231-41. doi: 10.11607/ofph.1413. PMID 26244431
- [Background] Costa YM, Porporatti AL, Stuginski-Barbosa J, Bonjardim LR, Conti PC. Additional effect of occlusal splints on the improvement of psychological aspects in temporomandibular disorder subjects: A randomized controlled trial. Arch Oral Biol. 2015 May;60(5):738-44. doi: 10.1016/j.archoralbio.2015.02.005. Epub 2015 Feb 20. PMID 25768709
- [Background] Jacobson E. Interview with Edmund Jacobson. Biofeedback Self Regul. 1978 Sep;3(3):287-300. doi: 10.1007/BF00999297. No abstract available. PMID 728486
- [Background] Golombek U. [Progressive muscle relaxation (PMR) according to Jacobson in a department of psychiatry and psychotherapy - empirical results]. Psychiatr Prax. 2001 Nov;28(8):402-4. doi: 10.1055/s-2001-18615. German. PMID 11721228
- [Background] Wilk C, Turkoski B. Progressive muscle relaxation in cardiac rehabilitation: a pilot study. Rehabil Nurs. 2001 Nov-Dec;26(6):238-42; discussion 243. doi: 10.1002/j.2048-7940.2001.tb01963.x. PMID 12035725
- [Background] Grossi ML, Goldberg MB, Locker D, Tenenbaum HC. Irritable bowel syndrome patients versus responding and nonresponding temporomandibular disorder patients: a neuropsychologic profile comparative study. Int J Prosthodont. 2008 May-Jun;21(3):201-9. PMID 18548956
- [Background] Takemura T, Takahashi T, Fukuda M, Ohnuki T, Asunuma T, Masuda Y, Kondoh H, Kanbayashi T, Shimizu T. A psychological study on patients with masticatory muscle disorder and sleep bruxism. Cranio. 2006 Jul;24(3):191-6. doi: 10.1179/crn.2006.031. PMID 16933460
- [Background] van Selms MK, Lobbezoo F, Visscher CM, Naeije M. Myofascial temporomandibular disorder pain, parafunctions and psychological stress. J Oral Rehabil. 2008 Jan;35(1):45-52. doi: 10.1111/j.1365-2842.2007.01795.x. PMID 18190360
- [Background] Hutchings DF, Reinking RH. Tension headaches: what form of therapy is most effective? Biofeedback Self Regul. 1976 Jun;1(2):183-90. doi: 10.1007/BF00998585. PMID 791381
- See also: Incidence of temporomandibular disorders - parafunctions and dysfunctions in dental students - the comparative studies — http://www.czytelniamedyczna.pl/1776,ocena-czestosci-wystepowania-zaburzen-czynnosciowych-narzadu-zucia-w-grupie-stud.html
- See also: Influence of Selected Psychoemotional Factors on the Prevalence of Bruxism — http://www.dbc.wroc.pl/Content/1892/DMP_2006431089_Mank.pdf